CLINICAL TRIAL: NCT00550108
Title: A Prospective Study of the Management of Incidentally Discovered Pancreatic Cysts
Brief Title: Management of Incidentally Discovered Pancreatic Cysts
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to enroll subjects.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Cristina R. Ferrone, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-P-000420
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Pancreatic Cyst
Keywords: pancreatic cyst; ethanol injection
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Observation of pancreatic cysts
- B (Experimental): Ethanol lavage of pancreatic cysts
  Interventions: Other: Ethanol lavage

INTERVENTIONS:
Other: Ethanol lavage — Ethanol lavage of pancreatic cysts.
  Arms: B

SUMMARY:
The purpose of this study is to determine the natural history of pancreatic cysts and to determine if these cysts can be effectively treated with a less invasive therapy (ethanol injection vs periodic imaging) rather than surgical resection

DETAILED DESCRIPTION:
The appropriate management of patients with cystic lesions of the pancreas is controversial. The identification of small asymptomatic pancreatic cysts is increasing due to an improvement in the quality of radiologic imaging and the frequency that imaging is obtained. However, the natural history of these lesions is unknown1. The current consensus guidelines established at the International Consensus Conference in Sendai, Japan in 2005 suggest that branch chain IPMNs and mucinous cystic neoplasms that cause no symptoms, measure <3cm, and have no nodules can be observed with periodic imaging. However, the time course of these pre malignant mucinous lesions, intraductal papillary mucinous neoplasms (IPMN) or mucinous cystadenomas, from benign to malignant has not been determined. Due to the unknown natural history, and diagnostic uncertainty, some authors have recommended routine resection2, 3. Resection, despite improvements in surgical outcomes after pancreatectomy at high volume centers, carries a mortality and morbidity of 1-6% and 35-51%, respectively4-6. More recently studies are reporting a more selective approach to avoid the risk of operation in patients with benign lesions7. Improved radiographic and endoscopic studies have been able to identify some lesions with increased malignant potential8, 9. Thus, most patients will undergo pancreas specific radiologic imaging and endoscopic ultrasound with cyst aspiration. Since the natural history of cystic lesions is poorly understood no clear guidelines for surgical resection have been established. Some of the cysts will grow over time, with an increase in the cumulative risk of malignancy. Therefore, the therapeutic alternatives are to wait and watch for a change in the cyst morphology or to treat preemptively, which has been restricted to surgical resection. Based on the pilot study performed by Dr. William Brugge, at Massachusetts General Hospital, ethanol lavage of pancreatic cysts is safe and will result in a decrease in cyst diameter in 61% of patients. Additionally, if patients elect to not be treated preemptively it is unclear how to best follow these patients in terms of the type and the frequency of follow up studies.

ELIGIBILITY:
Inclusion Criteria:

* Cyst between 1-3cm
* No evidence of a mural nodule, solid component, or septations in the cyst
* For patients with multiple cysts, the largest will be evaluated

Exclusion Criteria:

* Any imaging or cytology concerning for malignancy
* Pancreatic Pseudocyst
* Gross Cyst >3cm as measured on MRCP
* Clinically active pancreatitis or serum amylase or lipase >3x upper limit of normal
* Coagulopathy (INR>1.5, PTT>100, Platelets<50K)
* Inability to tolerate conscious sedation and endoscopy
* Rated ASA IV or greater
* Prior EUS and aspiration of the pancreatic cyst
* Breast feeding
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Patients not progressing to operation due to the development of symptoms, growth to a maximum diameter of >3cm, or development of a mural nodule. | 3 years

SECONDARY OUTCOMES:
A decrease in size by >1 cm on MRCP Relative decrease in size of cyst after 1 or 2 injections with ethanol Is reduction in size durable (over what length of time)? | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina R Ferrone, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fernandez-del Castillo C, Targarona J, Thayer SP, Rattner DW, Brugge WR, Warshaw AL. Incidental pancreatic cysts: clinicopathologic characteristics and comparison with symptomatic patients. Arch Surg. 2003 Apr;138(4):427-3; discussion 433-4. doi: 10.1001/archsurg.138.4.427. PMID 12686529